CLINICAL TRIAL: NCT00742274
Title: A Randomized European Study Comparing Endoluminal Stent Grafting and Best Medical Therapy (BMT) to BMT Alone in the Treatment of Acute Uncomplicated Type B Aortic Dissection
Brief Title: A European Study on Medical Management Versus TAG Device + Medical Management for Acute Uncomplicated Type B Dissection
Acronym: ADSORB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAG 05-04
Record Dates: First submitted 2008-08-25; First posted 2008-08-27 (Estimated); Results first posted 2013-05-09 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-11

CONDITIONS: Aortic Diseases
MeSH Terms: conditions — Aortic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TAG+BMT
  Interventions: Device: Gore TAG Endoprosthesis
- 2 (Active Comparator): BMT alone
  Interventions: Other: Best Medical Therapy

INTERVENTIONS:
Device: Gore TAG Endoprosthesis — Implant Gore TAG device with Best Medical therapy per physician discretion
  Arms: 1
Other: Best Medical Therapy — Best Medical therapy is regimen of antihypertensive medications used to maintain blood pressure below 125/80 mm/Hg throughout the entire follow-up period. Because BMT is assessed by blood pressure response to medication, specific medication regimens for each patient will differ. The typical regimen consists of 1 to 4 concomitant antihypertensive medications that may include angiotensin converting enzyme (ACE) inhibitors, alpha blockers, beta blockers, calcium channel blockers, diuretics, and/or vasodilators.
  Arms: 2

SUMMARY:
The purpose of this study is to compare endoluminal stent grafting with the GORE TAG device and Best Medical Therapy (BMT) to BMT alone in the treatment of acute uncomplicated type B aortic dissections.

DETAILED DESCRIPTION:
Dissection of the aorta is a medical emergency requiring immediate surgery. Type B dissections are typically treated with surgery or endoluminal therapy when complications such as uncontrollable pain, organ ischemia, or aortic rupture are present. However, the treatment of patients with uncomplicated, acute type B dissections is controversial. Best medical therapy (BMT) is the standard of care in these cases since surgical repair offers no additional survival advantage. However, Endoluminal stent graft therapy with the GORE TAG Thoracic Endoprosthesis (GORE TAG device) may offer distinct advantages as an adjunct to medical therapy for uncomplicated acute type B dissection. The goal of endoluminal stent grafting is to cover the primary entry tear of the dissection to isolate the false lumen from blood flow and induce aortic remodeling.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of acute uncomplicated type B aortic dissection
2. Able to tolerate endotracheal intubation and general anesthesia
3. Maximum transverse diameter of the descending thoracic aorta < 55 mm and absence of descending thoracic aortic aneurysm, regardless of etiology.
4. Arterial anatomy is appropriate for stent graft therapy

Exclusion Criteria:

1. ASA classification = V
2. Severe renal insufficiency defined as SVS risk renal status = 3
3. Severe respiratory insufficiency defined as SVS risk pulmonary status = 3
4. Presence of connective tissue disease
5. Active infection or active vasculitides
6. Positive pregnancy test
7. Participation in another medical research study within 3 months of study enrollment
8. Myocardial infarction or cerebrovascular accident within 6 weeks prior to study enrollment
9. Planned concomitant surgical procedures (other than left subclavian artery transposition or bypass), or major surgery within 30 days of study enrollment
10. History of drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-08; Primary Completion 2012-02 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Brunkwall, MD, PhD, Principal Investigator — Kilinkum der Universitat zu Koln

REFERENCES:
- [Derived] Brunkwall J, Kasprzak P, Verhoeven E, Heijmen R, Taylor P; ADSORB Trialists; Alric P, Canaud L, Janotta M, Raithel D, Malina W, Resch T, Eckstein HH, Ockert S, Larzon T, Carlsson F, Schumacher H, Classen S, Schaub P, Lammer J, Lonn L, Clough RE, Rampoldi V, Trimarchi S, Fabiani JN, Bockler D, Kotelis D, Bockler D, Kotelis D, von Tenng-Kobligk H, Mangialardi N, Ronchey S, Dialetto G, Matoussevitch V. Endovascular repair of acute uncomplicated aortic type B dissection promotes aortic remodelling: 1 year results of the ADSORB trial. Eur J Vasc Endovasc Surg. 2014 Sep;48(3):285-91. doi: 10.1016/j.ejvs.2014.05.012. Epub 2014 Jun 22. PMID 24962744

RESULTS

PARTICIPANT FLOW:
Groups:
- TAG Device + Best Medical Therapy (BMT): TAG+BMT
- Best Medical Therapy (BMT) Alone: BMT alone
Period: Overall Study
Arm/Group | TAG Device + Best Medical Therapy (BMT) | Best Medical Therapy (BMT) Alone
Started | 30 | 31
Completed | 27 | 28
Not Completed | 3 | 3
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Removed for medical reasons | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TAG Device + Best Medical Therapy (BMT) | BEST MEDICAL THERAPY (BMT) Alone | Total
Number analyzed (Participants) | 30 | 31 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 19 | 36
  >=65 years | 13 | 12 | 25
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (10.5) | 60.7 (13.4) | 60.4 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 4 | 13
  Male | 21 | 27 | 48
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 0 | 1
  Denmark | 1 | 0 | 1
  France | 7 | 3 | 10
  Germany | 14 | 17 | 31
  Italy | 2 | 2 | 4
  Netherlands | 3 | 3 | 6
  Sweden | 1 | 4 | 5
  United Kingdom | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Composite of Partial or No False Lumen Thrombosis, Aortic Rupture, and Aortic Dilatation
Description: Subjects with any of the following met this composite outcome:
  * partial/no false lumen thrombosis
  * aortic rupture
  * aortic dilatation
  * lack of 1 year imaging (no image, incomplete image missing primary endpoint measurements, unevaluable image)
Time Frame: 1 year
Population: Intent to Treat (ITT)
Measure: Number; unit: participants
Arm/Group | TAG Device + Best Medical Therapy (BMT) | BEST MEDICAL THERAPY (BMT) Alone
Number analyzed (Participants) | 30 | 31
participants | 15 | 31
Statistical Analysis 1: Comparison: TAG Device + Best Medical Therapy (BMT) vs BEST MEDICAL THERAPY (BMT) Alone; Test type: Superiority or Other; p < 0.001, Chi-squared

ADVERSE EVENTS:
Arm/Group | TAG Device + Best Medical Therapy (BMT) | BEST MEDICAL THERAPY (BMT) Alone
Serious Adverse Events (participants affected / at risk) | 16/30 | 13/31
Other Adverse Events (participants affected / at risk) | 19/30 | 14/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAG Device + Best Medical Therapy (BMT) (N=30) | BEST MEDICAL THERAPY (BMT) Alone (N=31)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Mesenteric vascular insufficiency (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Death (General disorders) | 1 | 0
Device deployment issue (General disorders) | 2 | 0
Stent malfunction (General disorders) | 2 | 0
Stent-graft endoleak (General disorders) | 1 | 0
Hydrocholecystis (Hepatobiliary disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin T increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery dissection (Nervous system disorders) | 1 | 0
Paraplegia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Bronchopneumopathy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urostomy (Surgical and medical procedures) | 1 | 0
Aortic dilatation (Vascular disorders) | 2 | 4
Aortic dissection (Vascular disorders) | 0 | 1
Aortic intramural haematoma (Vascular disorders) | 0 | 1
Collateral circulation (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TAG Device + Best Medical Therapy (BMT) (N=30) | BEST MEDICAL THERAPY (BMT) Alone (N=31)
Angina pectoris (Cardiac disorders) | 3 | 2
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 2 | 0
Stent-graft endoleak (General disorders) | 2 | 0
Blood pressure abnormal (Investigations) | 7 | 4
Blood pressure increased (Investigations) | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Hypertension (Vascular disorders) | 5 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No